CLINICAL TRIAL: NCT05190822
Title: Evaluation of University Students' Knowledge Levels and Perceptions of the Physiotherapist in Turkey: A Health-Areas University Example
Brief Title: Evaluation of University Students' Knowledge Levels and Perceptions of the Physiotherapist
Status: Completed | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc Prof. Nuray Alaca, Acibadem University
Other Study IDs: ATADEK-2020-01/19
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Physical Therapist

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students
  Interventions: Other: College student

INTERVENTIONS:
Other: College student — Our research will be conducted by face-to-face interviews within the scope of questionnaires prepared by us for students studying in departments other than Physiotherapy and Rehabilitation at Acibadem Mehmet Ali Aydinlar University.

SUMMARY:
The aim of this study is to determine the knowledge, perceptions and perspectives of students about physiotherapy and rehabilitation profession, who are studying in different departments, especially in the health sector in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-25 who are students and continue their education at Acibadem Mehmet Ali Aydinlar University

Exclusion Criteria:

* Students in the physiotherapy and rehabilitation department
* Students with serious mental illness

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The current study will be conducted by face-to-face interviews within the scope of questionnaires prepared by us for students studying in departments other than Physiotherapy and Rehabilitation at Acibadem Mehmet Ali Aydinlar University
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of students about the physiotherapist profession | Baseline time
  5-point Likert (5=Strongly Agree, 0=Strongly Disagree) given to open-ended questions. As the score increases, the level of knowledge good [the minimum (18 point) and maximum values (90 point)], higher scores were mean a better outcome.
Perceptions of students about the physiotherapist profession | Baseline time
  Measuring perceptions of physiotherapist and other professions relative to each other (0-10). low scores indicate poor perception, high scores indicate good perception. [the minimum (8 point) and maximum values (80 point)], higher scores were mean a better outcome.

SECONDARY OUTCOMES:
Knowledge of students about the physiotherapist of health fields | Baseline time
  In which health fields does the physiotherapist profession work. As the number increases, the level of knowledge will be determined as good, as it decreases, it will be determined as bad. [the minimum (0 point) and maximum values (24 point)], higher scores were mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ALACA, Asocc. Prof, Study Director — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided